CLINICAL TRIAL: NCT06694467
Title: Improving Self-Efficacy, Quality of Life and Glycemic Control in Adolescents With Type 1 Diabetes: An Experimental Evaluation of the Family Centered Empowerment Model
Brief Title: Improving Self-Efficacy, Quality of Life and Glycemic Control in Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Salah Alzawahreh, RN, MSc, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU/2023/110-1681
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes mellitus; Quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): An official diabetes education program and family empowerment model where employed, designed to provide people with diabetes and their families the information and abilities they need to manage their condition effectively. Types of diabetes, blood sugar control, self-monitoring methods, nutrition, meal planning, physical activity recommendations, medication management, and problem-solving approaches are all included in these programs
  Interventions: Behavioral: Education program
- Control group (No Intervention): Patients diagnosed with type 1 diabetes mellitus for six months or more and had not attended any form of structured diabetes education including hospital-based classes or community group diabetes education classes for the preceding month of the study. These parameters were adopted to ensure that study takes place in a controlled environment and targets the aspects of intervention of study.

INTERVENTIONS:
Behavioral: Education program — An official diabetes education program designed to provide people with diabetes and their families the information and abilities they need to manage their condition effectively. Diabetes kinds, blood sugar control, self-monitoring methods, nutrition, meal planning, physical activity recommendations, medication management, and problem-solving approaches are all included in these programs. Additionally, they offer psychological assistance to help people manage the emotional challenges of having diabetes.
  Other Names: Diabetes education program
  Arms: Intervention group

SUMMARY:
Empowerment in healthcare, particularly in the context of chronic illness management such as diabetes, entails equipping patients with knowledge, expertise, and self-assurance to proactively oversee their health and make well-informed choices. This encompasses comprehensive strategies that target psychological, social, and lifestyle elements with the goal of enhancing self-confidence and health results. The objective of this research is to evaluate how the Family-Centered Empowerment Model affects the clinical and psychological outcomes of adolescents with Type 1 Diabetes, with an emphasis on increases in quality of life, self-efficacy, and glycosylated hemoglobin (HbA1c) levels.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a prevalent and increasingly acknowledged medical disorder that affects individuals worldwide. It is a metabolic condition marked by elevated blood glucose levels that can cause serious side effects like renal failure, heart disease, blindness, and even amputations. To provide a better understanding of the Family-Centered Empowerment Model intervention applied in this work, the components and delivery modes are described in more detail below. Furthermore, a figure or a table suggested at this part could help to present this information more shortly. Details about the intervention The Family-Centered Empowerment Model intervention aimed to help engage the adolescent, an individual with type 1 DM, and his/her family in the self management process. The purpose of this study was to improve coping skills with type 1 DM population by increasing teamwork between adolescents and their members of their household.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with type 1 diabetes, ages 12 to 18 years
* Patients who had not taken part in any professional diabetes education program within a month of receiving their diagnosis
* Patients who had been diagnosed at least six months earlier to the commencement of the study.

Exclusion Criteria:

* Adolescents who had severe long-term diseases
* Patients newly diagnosed type 1 diabetes.
* those who were enrolled in a diabetes education program one month or less prior to the commencement of the study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin level | 6 months
  Serum glycosylated hemoglobin level was measured as a baseline, then 6 months after the intervention, to measure the mean difference between the two readings.
Quality of life | 6 months
  Pediatric Quality of Life-Diabetes Module was used. The twenty-eight items in this multidimensional tool are categorized into five domains: treatment obstacles (four items), treatment adherence (seven items), concern (three items), and diabetic symptoms (eleven items). For teenage self-report, a five-point Likert scale was employed. The total number of questions divided by the total number of answers is how scale scores are calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Nicosia, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The study protocol, methodology, results, and the accompanying data will be published online after peer review process by the scientific journal to which it will be submitted.

REFERENCES:
- [Derived] Alzawahreh S, Ozturk C. Improving Self-Efficacy, Quality of Life, and Glycemic Control in Adolescents With Type 1 Diabetes: Randomized Controlled Trial for the Evaluation of the Family-Centered Empowerment Model. JMIR Form Res. 2024 Dec 10;8:e64463. doi: 10.2196/64463. PMID 39658013